CLINICAL TRIAL: NCT05491304
Title: Clinical Study on the Treatment of Pediatric Hemophagocytic Lymphohistiocytosis Based on Cytokine Guided Risk Stratification：A Multicenter Randomized Controlled Study
Brief Title: Cytokine Guided Risk Stratification and Treatment in Pediatric Hemophagocytic Lymphohistiocytosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Collaborators: The Second Hospital of Anhui Medical University (Other); Union hospital of Fujian Medical University (Other); Children's Hospital of Fudan University (Other); Zunyi Medical College (Other); Hunan Provincial People's Hospital (Other); Tongji Hospital (Other); Children's Hospital of Nanjing Medical University (Other); The Affiliated Hospital of Qingdao University (Other); Qilu Hospital of Shandong University (Other); Shanghai Children's Medical Center (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai Children's Hospital (Other); Shenzhen Children's Hospital (Other Government); West China Second University Hospital (Other); Children's Hospital of Soochow University (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Wuhan Children's Hospital (Other); Institute of Hematology & Blood Diseases Hospital, China (Other); The Third Xiangya Hospital of Central South University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xiaojun Xu, chief physician, The Children's Hospital of Zhejiang University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-IRB-057
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Hemophagocytic Lymphohistiocytoses; Cytokine Storm
Keywords: Hemophagocytic Lymphohistiocytoses; Cytokine Storm; Ruxolitinib; Interferon-gamma; Interleukin-10; Child; Stratification therapy
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic; Cytokine Release Syndrome | interventions — Dexamethasone; Steroids; Adrenal Cortex Hormones; Etoposide; ruxolitinib

STUDY DESIGN:
Intervention Model Description: The patients will be divide into different risk groups according to cytokine concentration, clinical manifestation and laboratory findings. For low/intermediate risk and not severe patients, steroid or ruxolitinib will be used initially; while those with high risk or "severe" disease, DXM+VP16±ruxolitinib will be administered.
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Non-severe DXM group (Experimental): Dexamethasone (DXM): week1-2: 10 mg/m2.d, week 3-4: 5 mg/m2.d, week5-6: 2.5 mg/m2.d, week7: 1.25 mg/m2.d, week8: tapering.
  Interventions: Drug: Dexamethasone
- Non-severe Ruxo group (Experimental): Ruxolitinib(Ruxo): body weight (BW)<10kg: 2.5mg Bid; 10-20kg: 5mg Bid; >20kg: 10mg Bid; Orally for 4 weeks.
  Interventions: Drug: Ruxolitinib
- Severe HLH-94 group (Experimental): DXM: week1-2: 10 mg/m2.d, week 3-4: 5 mg/m2.d, week5-6: 2.5 mg/m2.d, week7: 1.25 mg/m2.d, week8: tapering.
  Etoposide (VP16): 100-150mg/m2 twice in the first two weeks, and once every week to week 8.
  Interventions: Drug: Dexamethasone; Drug: Etoposide
- Severe HLH-94 plus ruxolitinib group (Experimental): DXM: week1-2: 10 mg/m2.d, week 3-4: 5 mg/m2.d, week5-6: 2.5 mg/m2.d, week7: 1.25 mg/m2.d, week8: tapering.
  Etoposide (VP16): 100-150mg/m2 twice in the first two weeks, and once every week to week 8.
  Ruxolitinib(Ruxo): body weight (BW)<10kg: 2.5mg Bid; 10-20kg: 5mg Bid; >20kg: 10mg Bid; Orally for 4 weeks.
  Interventions: Drug: Dexamethasone; Drug: Etoposide; Drug: Ruxolitinib

INTERVENTIONS:
Drug: Dexamethasone — Single drug in non-severe group; combined with etoposide±ruxolitinib in severe group.
  Other Names: Steroid; Corticosteroid
  Arms: Non-severe DXM group; Severe HLH-94 group; Severe HLH-94 plus ruxolitinib group
Drug: Etoposide — Used in severe group combined with etoposide.
  Other Names: VP16
  Arms: Severe HLH-94 group; Severe HLH-94 plus ruxolitinib group
Drug: Ruxolitinib — Single drug in non-severe group; combined with etoposide and dexamethasone in severe group.
  Other Names: JAK1/2 inhibitor
  Arms: Non-severe Ruxo group; Severe HLH-94 plus ruxolitinib group

SUMMARY:
Hemophagocytic lymphohistiocytosis (HLH) is a rapidly fatal disease caused by immune-dysregulation characterized by hypercytokinemia, with about 30%-40% of patients suffering death in children. Stratification strategy and individualized treatment is important to improve the survival. In our recent retrospective study, risk stratification based on IL-10 and IFN-γ levels well distinguished patients with different outcomes. In this multicenter prospective study, we will enroll the newly diagnosed pediatric HLH patients and divide them into low, intermediate and high-risk cytokine groups according to IFN-γ and IL-10 levels. The patients'clinical manifestation and laboratory findings will be further evaluated into severe and non-severe groups. For low/intermediate risk and non-severe patients, steroid or ruxolitinib will be used initially; while those with high risk or severe diseases, DXM+VP16±ruxolitinib will be administered. The treatment strategy could be adjusted after evaluation 48-72 hours later.

DETAILED DESCRIPTION:
Background and objectives: Hemophagocytic lymphohistiocytosis (HLH) is a rapidly fatal disease caused by immune-dysregulation characterized by hypercytokinemia, with about 30%-40% of patients suffering death in children. Early death is an important issue in HLH treatment, which is greatly caused by hypercytokinemia resulting in multi-organ disfunction and partially due to the treatment toxicities. Thus, stratification strategy and individualized treatment is important to improve the survival. In our recent retrospective study which enrolled 256 pediatric patients, the patients were stratified into low, intermediate and high risk according to their IL-10 and IFN-γ levels. The 8-week mortality for low, intermediate and high-risk patients were 5.4±2.4%, 16.9±3.4% and 48.7±8.0%, and the 5-year OS rate were 82.9±40%, 67.0±4.3% and 51.3±8.0%, respectively. This indicated that IFN-γ and IL-10 are helpful for stratifying HLH patients into different risk groups to receive individualized therapies. However, evidence of cytokine application based on multi-center prospective study is still lacking. The aim of this protocol is to establish a model to early identify the patients with low and high mortality and to guide the precise treatment of pediatric HLH.

Methods and protocol design: A multicenter prospective study in Asian countries is to be launched for children with HLH. The inclusion criterion is newly diagnosed pediatric HLH patients who has not received steroids or etoposide when enrollment. In this study, the patients are identified as low, intermediate and high-risk cytokine groups according to their cytokine levels: (1) low-risk: IFN-γ<3700pg/mL and IL-10<200pg/mL; (2) intermediate-risk: IFN-γ<3700pg/mL and IL-10≥200pg/mL; (3) high-risk: IFN-γ≥3700pg/mL. The patients' clinical manifestation and laboratory findings were evaluated as well and those fulfill either one of the following criteria were considered as "severe": (1) present ≥2 out of 3 ⅰ, albumin<26.0 g/L; ⅱ, direct bilirubin>55.0μmol/L; ⅲ, fibrinogen<0.75g/L. (2) CNS involvement, shock, mechanical ventilation, renal failure.

Based on the cytokine risk and disease severity, different intensity of treatment will be started. For low/intermediate risk and not severe patients, steroid or ruxolitinib will be used initially; while those with high risk or "severe" disease, DXM+VP16±ruxolitinib will be administered. The treatment strategy could be adjusted after evaluation 48-72 hours later based on treatment respose and cytokine levels. A total of 400 pediatric patients under 18 years old are to be recruited. The primary end-point of the study is the 8-week responsive rates and mortality, and one-year overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Age from one day to 18 years old；
* Newly diagnosed HLH, fulfilling the HLH criteria;
* To observed the early diagnosis role of cytokines, patients who is suspected to be HLH and fulfill 3 out of 8 criteria can be pre-enrolled.

Exclusion Criteria:

* treated with steroids or etoposide within 72 hours before diagnosis.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete remission (CR) | 8th week after the initial of therapy
  Complete remission rate in 8th week
Overall survival (OS) | One year after enrollment
  Overall survival rate in one year
overall response rate (ORR) | At the 4th and 8th week of treatment
  including the proportion of patients achieving CR, PR and HLH improvement
Mortality | At the 8th week of diagnosis
  8-week mortality

SECONDARY OUTCOMES:
Reactivation rate | Any time during the first year after diagnosis
  The relapse rate of disease
Partial remission (PR) | 4th week after the initial of therapy
  Partial remission rate in 4th week
Rate of Early Death | 2nd week after diagnosis
  Death occurred within 2 weeks after diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Xu, MD, Principal Investigator — The Children's Hospital of Zhejiang University School of Medicine; Yongmin Tang, MD, Principal Investigator — The Children's Hospital of Zhejiang University School of Medicine
Locations (1):
- The Children's Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bergsten E, Horne A, Arico M, Astigarraga I, Egeler RM, Filipovich AH, Ishii E, Janka G, Ladisch S, Lehmberg K, McClain KL, Minkov M, Montgomery S, Nanduri V, Rosso D, Henter JI. Confirmed efficacy of etoposide and dexamethasone in HLH treatment: long-term results of the cooperative HLH-2004 study. Blood. 2017 Dec 21;130(25):2728-2738. doi: 10.1182/blood-2017-06-788349. Epub 2017 Sep 21. PMID 28935695
- [Background] Xu XJ, Tang YM. Dilemmas in diagnosis and management of hemophagocytic lymphohistiocytosis in children. World J Pediatr. 2020 Aug;16(4):333-340. doi: 10.1007/s12519-019-00299-3. Epub 2019 Sep 10. PMID 31506890
- [Background] Tang Y, Xu X, Song H, Yang S, Shi S, Wei J, Pan B, Zhao F, Liao C, Luo C. Early diagnostic and prognostic significance of a specific Th1/Th2 cytokine pattern in children with haemophagocytic syndrome. Br J Haematol. 2008 Oct;143(1):84-91. doi: 10.1111/j.1365-2141.2008.07298.x. Epub 2008 Jul 31. PMID 18673367
- [Background] Xu XJ, Tang YM, Song H, Yang SL, Xu WQ, Zhao N, Shi SW, Shen HP, Mao JQ, Zhang LY, Pan BH. Diagnostic accuracy of a specific cytokine pattern in hemophagocytic lymphohistiocytosis in children. J Pediatr. 2012 Jun;160(6):984-90.e1. doi: 10.1016/j.jpeds.2011.11.046. Epub 2012 Jan 9. PMID 22226576
- [Background] Xu XJ, Luo ZB, Song H, Xu WQ, Henter JI, Zhao N, Wu MH, Tang YM. Simple Evaluation of Clinical Situation and Subtypes of Pediatric Hemophagocytic Lymphohistiocytosis by Cytokine Patterns. Front Immunol. 2022 Feb 28;13:850443. doi: 10.3389/fimmu.2022.850443. eCollection 2022. PMID 35296096
- [Background] Wang J, Zhang R, Wu X, Li F, Yang H, Liu L, Guo H, Zhang X, Mai H, Li H, Wang Z. Ruxolitinib-combined doxorubicin-etoposide-methylprednisolone regimen as a salvage therapy for refractory/relapsed haemophagocytic lymphohistiocytosis: a single-arm, multicentre, phase 2 trial. Br J Haematol. 2021 May;193(4):761-768. doi: 10.1111/bjh.17331. Epub 2021 Feb 9. PMID 33559893
- [Background] Zhang Q, Zhao YZ, Ma HH, Wang D, Cui L, Li WJ, Wei A, Wang CJ, Wang TY, Li ZG, Zhang R. A study of ruxolitinib response-based stratified treatment for pediatric hemophagocytic lymphohistiocytosis. Blood. 2022 Jun 16;139(24):3493-3504. doi: 10.1182/blood.2021014860. PMID 35344583
- [Background] Ehl S, Astigarraga I, von Bahr Greenwood T, Hines M, Horne A, Ishii E, Janka G, Jordan MB, La Rosee P, Lehmberg K, Machowicz R, Nichols KE, Sieni E, Wang Z, Henter JI. Recommendations for the Use of Etoposide-Based Therapy and Bone Marrow Transplantation for the Treatment of HLH: Consensus Statements by the HLH Steering Committee of the Histiocyte Society. J Allergy Clin Immunol Pract. 2018 Sep-Oct;6(5):1508-1517. doi: 10.1016/j.jaip.2018.05.031. Epub 2018 Jul 4. PMID 30201097
- [Background] Henter JI, Horne A, Arico M, Egeler RM, Filipovich AH, Imashuku S, Ladisch S, McClain K, Webb D, Winiarski J, Janka G. HLH-2004: Diagnostic and therapeutic guidelines for hemophagocytic lymphohistiocytosis. Pediatr Blood Cancer. 2007 Feb;48(2):124-31. doi: 10.1002/pbc.21039. PMID 16937360